CLINICAL TRIAL: NCT06522113
Title: Cilostazol and Aspirin in Acute Minor Stroke and Transient Ischemic Attack
Brief Title: Cilostazol and Aspirin in Stroke and TIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Incheon St.Mary's Hospital (Other)
Responsible Party: Principal Investigator, Taewon Kim, Principal Investigator, Incheon St.Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OC23RISI0149
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Ischemic Stroke; TIA
MeSH Terms: conditions — Ischemic Stroke | interventions — Cilostazol; Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aspirin with clopidogrel (Active Comparator): aspirin 100mg with clopidogrel 75mg for 21 days
  Interventions: Drug: Clopidogrel
- aspirin with cilostazol (Experimental): aspirin 100mg with cilostazol 200 mg for 21 days
  Interventions: Drug: Cilostazol

INTERVENTIONS:
Drug: Cilostazol — patients were given cilostazol 100mg twice a day with aspirin
  Other Names: aspirin
  Arms: aspirin with cilostazol
Drug: Clopidogrel — patients were given clopidogrel 75mg with aspirin
  Other Names: aspirin
  Arms: aspirin with clopidogrel

SUMMARY:
This study is a randomized, open-labelled trial. We randomly assigned patients within 24 hours after the onset of minor ischemic stroke or high-risk TIA to combination therapy with cilostazol and aspirin or to clopidogrel plus aspirin. The primary outcome was stroke (ischemic or hemorrhagic) during 90 days of follow-up in an intention-to-treat analysis.

DETAILED DESCRIPTION:
This study is a randomized, open-labelled trial. We randomly assigned patients within 24 hours after the onset of minor ischemic stroke or high-risk TIA to combination therapy with cilostazol and aspirin (aspirin 100mg with cilostazol 200 mg for 21 days) or to clopidogrel plus aspirin (aspirin 100mg with clopidogrel 75mg for 21 days). The primary outcome was stroke (ischemic or hemorrhagic) during 90 days of follow-up in an intention-to-treat analysis. The primary safety outcome was the moderate-to-severe bleeding event according to (GUSTO) definition. The secondary outcomes were new clinical vascular event (ischemic or hemorrhagic stroke, myocardial infarction, or vascular death), analyzed as a composite outcome and also as individual outcomes. Vascular death was defined as death due to stroke (ischemic or hemorrhagic), systemic hemorrhage, myocardial infarction, congestive heart failure, pulmonary embolism, sudden death, or arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of an acute minor ischemic stroke or TIA
* Acute minor stroke was defined by a score of 3 or less at the time of randomization on the National Institutes of Health Stroke Scale (NIHSS; scores range from 0 to 42, with higher scores indicating greater deficits)

Exclusion Criteria:

* Intracerebral Hemorrhage
* Brain tumor
* Brain abscess, or other major non-ischemic brain disease;
* Isolated sensory symptoms (numbness, isolated visual changes, or isolated dizziness or vertigo) without evidence of acute infarction on baseline CT or MRI of the head
* A score of more than 2 on the modified Rankin scale, immediately before the occurrence of the index ischemic stroke or TIA, indicating moderate disability or worse at baseline
* An NIHSS score of 4 or more at randomization
* A clear indication for anticoagulation therapy (presumed cardiac source of embolus, such as atrial fibrillation or prosthetic cardiac valve) or a contraindication to clopidogrel, cilostazol or aspirin
* History of intracranial hemorrhage
* Anticipated requirement for long-term non-study antiplatelet drugs or for nonsteroidal anti-inflammatory drugs affecting platelet function
* Heparin therapy or oral anticoagulation therapy within 10 days before randomization
* Gastrointestinal bleeding or major surgery within the previous 3 months
* Planned or probable revascularization (any angioplasty or vascular surgery) within 3 months after screening (if clinically indicated, vascular imaging was to be performed before randomization, whenever possible)
* Planned surgery or interventional treatment requiring cessation of the study drug
* TIA or minor stroke caused by angiography or surgery
* Severe non- cardiovascular coexisting condition, with a life expectancy of less than 3 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
New stroke event for 90 days (Ischemic or hemorrhagic) | for 90 days
  New stroke event for 90 days (Ischemic or hemorrhagic)
Moderate-to-severe bleeding event according to (GUSTO) definition | for 90 days
  Moderate-to-severe bleeding event according to (GUSTO) definition:
  Moderate : bleeding requiring transfusion Severe : Fatal or intracerebral bleeding, or bleeding resulting in substantial hemodynamic compromise requiring treatment

SECONDARY OUTCOMES:
New clinical vascular event (ischemic or hemorrhagic stroke, myocardial infarction, or vascular death), analyzed as a composite outcome and also as individual outcomes. | for 90 days
  New clinical vascular event (ischemic or hemorrhagic stroke, myocardial infarction, or vascular death), analyzed as a composite outcome and also as individual outcomes. Vascular death was defined as death due to stroke (ischemic or hemorrhagic), systemic hemorrhage, myocardial infarction, congestive heart failure, pulmonary embolism, sudden death, or arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Taewon Kim, Dr, Principal Investigator — the catholic university of korea, neurology department
Locations (1):
- The Catholic university of korea, Incheon St. Mary's hospital, Incheon, South Korea